CLINICAL TRIAL: NCT06102083
Title: A Phase II, Multi-center, Randomized, Double-blinded, Placebo-controlled Clinical Study Evaluating the Efficacy and Safety of TDI01 Suspension for the Treatment of Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: A Clinical Trial on the Treatment of Idiopathic Pulmonary Fibrosis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Tide Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDI01-IPF-II-01
Record Dates: First submitted 2023-07-31; First posted 2023-10-26 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental group 1 (Experimental): TDI01 dose A, once daily
  Interventions: Drug: TDI01 suspension
- Experimental group 2 (Experimental): TDI01 dose B, once daily
  Interventions: Drug: TDI01 suspension
- Control group (Placebo Comparator): Placebo, once daily
  Interventions: Drug: TDI01 suspension

INTERVENTIONS:
Drug: TDI01 suspension — Experimental group 1:
  Drug: TDI01 suspension Administration: TDI01 suspension once daily.
  Experimental group 2:
  Drug: TDI01 suspension Administration: TDI01 suspension once daily.
  Control group:
  Drug: Placebo Administration: Placebo once daily.

SUMMARY:
This trial was performed in patients with idiopathic pulmonary fibrosis (IPF) to evaluate the clinical efficacy and safety of different doses of TDI01 Suspension, compared with control, for the treatment of patients with IPF.

DETAILED DESCRIPTION:
This is a Phase II, multi-center, randomized, double-blinded, placebo-controlled clinical study to evaluate the efficacy and safety of TDI01 Suspension for the treatment of IPF. The study consists of a 4-week screening period, a 24-week treatment period, a 28-week extension period, and a 2-week safety follow-up period.

It is planned to include 120 IPF patients. All subjects will be randomized in a 1:1:1 ratio to receive a 24-week treatment with TDI01 Suspension dosage A, TDI01 Suspension dosage B, or the placebo. At Week 24, the subjects will be evaluated for the primary efficacy endpoints and subsequently enter the extension period. Subjects may continue receiving the investigational product until Week 52 at their voluntary consent.

ELIGIBILITY:
Inclusion Criteria

1. Females or males aged 40 to 80 (inclusive) at the time of signing the ICF;
2. Is willing to participate voluntarily in this clinical study and sign the ICF prior to study initiation;
3. Diagnosed with Idiopathic Pulmonary Fibrosis (IPF) according to the principles of the 2022 ATS/ERS/JRS/ALAT clinical practice guidelines;
4. Females or males of reproductive potential must agree and commit to using effective contraception from the time of signing the ICF until 90 days after the last dose of the investigational product;
5. Has stable anti-fibrosis treatment for at least 12 weeks prior to Visit 1.
6. FEV1/FVC ≥0.70 at screening;
7. Percent predicted forced vital capacity (% FVC) ≥45% and ≤90% at screening;
8. DLco% (Hb corrected) ≥30% and ≤90% at screening;
9. Is willing and able to comply with the protocol and attend visits as assessed by the investigator.

Exclusion Criteria

Subjects are not eligible for participation in the study if they meet any of the following exclusion criteria:

1. Patients with interstitial lung disease caused by other known aetiology;
2. Patients who experienced active tuberculosis infection within 12 months prior to screening, or present any bacterial, viral, parasitic, or fungal infection requiring treatment at screening;
3. Patients with IPF significantly worsened within one month prior to randomization;
4. Patients with range of emphysema more than that of pulmonary fibrosis as indicated by chest HRCT at screening;
5. Patients who are expected to undergo a lung transplant during the course of the study or have an expected survival of less than 1 year;
6. Patients who received any of the following medications within 28 days prior to randomization, such as unstable anti-fibrosis treatment, >15 mg/d prednisone or equivalent dose of other glucocorticoids, immunomodulatory agents,strong inhibitors of CYP3A4;
7. Patients with a history of malignancy within 5 years prior to screening (except for patients with appropriately treated basal cell carcinoma of the skin or squamous cell carcinoma in situ of the skin or carcinoma in situ of the cervix);
8. Patients with moderate to severe hepatic insufficiency (Child-Pugh class B or C) prior to screening;
9. Patients with laboratory test results exceeding any of the following criteria at screening: total bilirubin >1.5 x ULN or AST/ALT >2 x ULN, and serum CK >2.5 x ULN;
10. Patients with uncontrolled hepatitis B virus infection or hepatitis C virus infection at screening;
11. Patients with a history of unstable or worsening cardiac disease within 6 months prior to screening;
12. Patients with a family or personal history of long QT syndrome or QTcF >480 ms at screening;
13. Patients with a creatinine clearance (CLcr) <50 mL/min at screening, calculated using the Cockcroft-Gault formula;
14. Patients who are unable to complete the 6MWD test or PFT;
15. Pregnant or lactating women; Further exclusion criteria apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-11-02 (Estimated); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Forced Vital Capacity (FVC) (mL) at Week 24 | At 24 week
  The mean change in FVC (ml) from baseline at week 24, measured by spirometer

SECONDARY OUTCOMES:
Change From Baseline in FVC% Predicted | From baseline up to week 52
  The change in FVC as a percentage of expected value (FVC%) ffrom baseline measured by spirometer.
  The time points which will be measured are from baseline to Week 12, Week 24, Extension Week 32, Extension Week 40, and Extension Week 52.
Proportion of Subjects with an Absolute Decrease of FVC% Predicted Greater than 10% | From baseline up to week 52
  The proportion of subjects with an absolute decrease of FVC% greater than 10% measured by spirometer from baseline. The time point which will be measured are from baseline to Week 24, and Extension Week 52.
Change From Baseline in Diffusing Capacity (of Lung) for Carbon Monoxide (DLCO) % | From baseline up to week 24
  The Change of DLCO% with Hb correction measured by spirometer from baseline. The time point which will be measured are from baseline to Week 12 and Week 24.
Time to First Acute Idiopathic Pulmonary Fibrosis (IPF) Exacerbation | From baseline up to week 52
  Time to first acute idiopathic pulmonary fibrosis exacerbation during the trial.
Time to Disease Progression | From baseline up to week 52
  Time to Disease Progression during the trial. Disease progression is defined as 10% absolute decrease in FVC, lung transplant or death, whichever occurs first.
Mean Change in Distance Walked in the 6-minute Walk Test (6MWT) | From baseline up to week 24
  The mean change in 6MWD. The time points which will be measured are from baseline to Week 12 and Week 24.
The change in St.George's respiratory questionnaire（SGRQ） | From baseline up to week 24
  The mean change in total score of SGRQ from basline to Week 12 and Week 24. The SGRQ is a standardized self-completed questionnaire for measuring impaired health and perceived well-being in airways disease. It consists of multiple parts on different scales related to each question to assess the impact of respiration on the subject's life.
  A total score is ranged from 0 (no health impairment) to 100 (maximum health impairment). The lower the better.